CLINICAL TRIAL: NCT03066232
Title: Delirium in Home-dwelling Old People Receiving Home Nursing Care
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Sandefjord kommune (Unknown); Norwegian Centre for Ageing and Health (Other); The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Maria Krogseth, MD, PhD, Oslo University Hospital
Other Study IDs: 2014/1972
Record Dates: First submitted 2017-02-20; First posted 2017-02-28 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Delirium
Keywords: Delirium; Dementia; Physical function
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the prevalence of delirium among old persons with home-nursing care living in the community. By recruiting the persons in a stable phase, the investigators wish to study the influence of an episode of delirium upon further cognitive and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Home nursing service at least once a week.
* Home dwelling (not permanently institutionalised)
* Age 65 years or more
* Informed consent by the patient or a close relative (if the patient is unable to give a valid informed consent)

Exclusion Criteria:

* Patient or relative denies inclusion
* Terminal illness
* Patients diagnosed with dementia with Lewy bodies (its fluctuating course makes the diagnosis of delirium challenging)
* Patients with chronic diseases that have needed assistance from the home nursing service before the age of 65.
* Assistance from the home nursing service is due to addictive substances.
* Assistance from the home nursing service is due to psychiatric illnesses other than dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Persons older than 65 years living in their own home receiving home nursing care at least once a week.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Trajectory of cognitive function using the MoCa test | 2 years
  The impact of an episode of delirium upon cognitive function measured by the Montreal Cognitive Assessment every 6th months for two years.

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Bruun Wyller, MD, PhD, Study Chair — Oslo University Hospital, University of Oslo
Locations (1):
- Sandefjord kommune, Sandefjord, Norway

IPD SHARING:
Plan to Share IPD: No